CLINICAL TRIAL: NCT00788749
Title: A Proof Of Concept Study to Investigate the Clinical, Histological And Molecular Predictors of Response to Oral and Intranasal Corticosteroid in Nasal Polyposis
Brief Title: Medical Polypectomy and Predictors of Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); NHS Tayside (Other Government)
Responsible Party: Sriram Vaidyanathan, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GRAY07
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Nasal Polyps
Keywords: chronic rhinosinusitis; nasal polyps; oral steroid; intranasal steroid; medical polypectomy
MeSH Terms: conditions — Nasal Polyps | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets for 2 weeks followed by fluticasone nasal drops 800mcg/d for 2 months followed by fluticasone nasal spray 400 mcg/d for 4 months
  Interventions: Drug: Placebo; Other: fluticasone nasal drops; Other: fluticasone nasal spray
- Prednisolone (Experimental): 25 mg Prednisolone OD for 2 weeks followed by Fluticasone nasal drops 800 mcg/d for 2 months, followed by fluticasone nasal spray 400mcg/day for 4 months
  Interventions: Drug: Prednisolone; Other: fluticasone nasal drops; Other: fluticasone nasal spray

INTERVENTIONS:
Drug: Prednisolone — tablets 25 mg/day
  Arms: Prednisolone
Drug: Placebo — tablets once daily
  Arms: Placebo
Other: fluticasone nasal drops — fluticasone nasal drops 800mcg/d
Other: fluticasone nasal spray — fluticasone nasal spray 400 mcg/d

SUMMARY:
This is the first randomized parallel group clinical trial looking at oral prednisolone induced medical nasal polypectomy followed by maintenance on topical steroid therapy in patients with nasal polyposis. This study also looks at the effect of aspirin sensitivity and the factors linking nasal polyps with asthma. We have also taken baseline measurements of a variety of blood, surface and biopsy markers to assess for potential to predict steroid response. Finally, the still unchartered link between nasal polyps and asthma will be explored by measuring Staphylococcal superantigens in serum before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 18-75 years of age
* bilateral nasal polyposis Grade 2 and above
* with or without asthma
* with or without atopy or aspirin sensitivity
* written informed consent

Exclusion Criteria:

* unilateral nasal polyposis
* polypoid lesion suspicious of inverted papilloma, malignancy, Wegeners granulomatosis, sarcoidosis
* known or suspected hypersensitivity to fluticasone propionate or any other constituents of the Investigational Medicinal product (IMP).
* Any clinically significant medical condition or abnormality, which, in the opinion of the investigator, might compromise the safety of the subject or which might interfere with the study.
* significant (≥50%)septal deviation
* inability to comply with the requirements of the protocol
* females who are pregnant, lactating or planning to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-05; Primary Completion 2008-02 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Endoscopy Polyp Grading | 0, 2 weeks, 10 weeks, 28 weeks

SECONDARY OUTCOMES:
Mini RQLQ | 0, 2 wks, 10 wks, 28 wks
TNS-4 | 0, 2 wks, 10 wks, 28 wks
PNIF | 0,2 wks, 10 wks,28 wks
Anosmia score | 0, 2 wks, 10 wks, 28 wks
Scratch n Sniff cards | 0, 2 wks, 10 wks, 28 wks
OUCC | 0, 2 wks, 10 wks, 28 wks
1 mcg Synacthen test | 0, 2 wks, 10 wks, 28 wks

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Vaidyanathan, MRCS, Principal Investigator — University of Dundee; Brian J Lipworth, MD, Study Director — University of Dundee
Locations (1):
- Ninewells Hospital and Medical School, Dundee, Angus, United Kingdom

REFERENCES:
- [Derived] Williamson PA, Vaidyanathan S, Clearie K, Barnes M, Lipworth BJ. Airway dysfunction in nasal polyposis: a spectrum of asthmatic disease? Clin Exp Allergy. 2011 Oct;41(10):1379-85. doi: 10.1111/j.1365-2222.2011.03793.x. Epub 2011 Jun 16. PMID 21676042
- [Derived] Vaidyanathan S, Barnes M, Williamson P, Hopkinson P, Donnan PT, Lipworth B. Treatment of chronic rhinosinusitis with nasal polyposis with oral steroids followed by topical steroids: a randomized trial. Ann Intern Med. 2011 Mar 1;154(5):293-302. doi: 10.7326/0003-4819-154-5-201103010-00003. PMID 21357906